CLINICAL TRIAL: NCT01129050
Title: Effects of Plant and Marine Omega-3 (w-3) Fatty Acids on Inflammatory Markers In Insulin Resistant Adults
Brief Title: Effects of Omega-3 Fatty Acids on Markers of Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Christopher Gardner, Professor of Medicine (Research), Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SU-05042010-5842; R21AT003465-01 (NIH)
Record Dates: First submitted 2010-05-20; First posted 2010-05-24 (Estimated); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Obesity; Hypertriglyceridemia; Insulin Resistance; Hypertension
Keywords: Fish oil; Omega-3 fatty acids; Metabolic syndrome; Adults
MeSH Terms: conditions — Obesity; Hypertriglyceridemia; Insulin Resistance; Hypertension; Metabolic Syndrome | interventions — Fish Oils; Linseed Oil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Low-dose Flaxseed Oil (Experimental): 2.2 g ALA (alpha-linolenic acid) per day
  Interventions: Dietary Supplement: Flaxseed Oil
- High-dose Flaxseed Oil (Experimental): 6.6 g ALA (alpha-linolenic acid) per day
  Interventions: Dietary Supplement: Flaxseed Oil
- Low-dose Fish Oil (Experimental): 1.2 g EPA+DHA (700 mg EPA and 500 mg DHA) per day
  Interventions: Dietary Supplement: Fish Oil
- High-dose Fish Oil (Experimental): 3.6 g EPA+DHA (2.1 g EPA and 1.5 g DHA) per day
  Interventions: Dietary Supplement: Fish Oil
- Placebo (Placebo Comparator): 4 g or 6 g soybean oil per day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fish Oil — Fish oil capsule
  Arms: High-dose Fish Oil; Low-dose Fish Oil
Dietary Supplement: Flaxseed Oil — Flaxseed oil capsule
  Arms: High-dose Flaxseed Oil; Low-dose Flaxseed Oil
Dietary Supplement: Placebo — Soybean oil capsule
  Arms: Placebo

SUMMARY:
The major purpose of this study is to examine the effect of two sources of dietary omega-3 fatty acids, each given at two doses, on potential health benefits related to cardiovascular disease prevention. The two sources of dietary omega-3 fatty acids will be fish oil, and flaxseed oil.

DETAILED DESCRIPTION:
The primary aim of this study is to examine the effect of two sources of dietary omega-3 fatty acids, each given at two doses, on potential health benefits related to cardiovascular disease prevention. The two sources of dietary omega-3 fatty acids will be fish oil, and flaxseed oil. Each will be given at a lower dose that could realistically be achieved from food sources alone, and at a higher dose that could not realistically be achieved from food alone and would require supplementation. The outcomes being studied are markers of inflammation. The subjects being studied are those with elevated risk factors for diabetes and heart disease that meet the criteria for the "metabolic syndrome". These are the people who are currently not diabetic, and who have not been diagnosed yet with heart disease, who are at risk of developing these diseases and who would likely benefit the most from the omega-3 therapy should it prove to be effective.

ELIGIBILITY:
Inclusion Criteria:Gender:

* Both women and men
* Age: > or = 18 years
* Ethnicity and race: All ethnic and racial backgrounds welcome
* As defined in ATP III of the National Cholesterol Education program, the metabolic syndrome will be diagnosed as presence of at least three of the following, which will be measured at the screening clinic visit:

Central obesity as measured by waist circumference:

* Men: Greater than 40 inches
* Women: Greater than 35 inches

  * Fasting blood triglycerides greater than or equal to 150 mg/dL
  * Blood HDL cholesterol:
* Men: Less than 40 mg/dL
* Women: Less than 50 mg/dL

  * Blood pressure greater than or equal to 130/85 mmHg

    * Fasting glucose greater than or equal to 100 mg/dL

Planning to be available for clinic visits and bottle pick-ups for the 8 weeks of study participation

Ability and willingness to give written informed consent

No known active psychiatric illness.

Exclusion Criteria:Daily intake of dietary supplements containing omega-3 FAs within the past month.

* Fasting blood glucose > 140 mg/dL
* Significant liver enzyme abnormality
* AST or ALT more than 2 times the upper limit of normal and/or
* Bilirubin more than 50% the upper limit of normal
* Renal disease as measured at baseline:
* Serum creatinine > 1.30 mg/dL, or
* Calculated creatinine clearance < 71 mL/min
* Self reported personal history of:

  * Clotting disorders
  * Clinically significant atherosclerosis (e.g., CAD, PAD)
  * Malignant neoplasm
  * Ongoing infection
  * Inflammatory disease (e.g., rheumatoid arthritis)
* Subjects currently receiving the following medications (self report):

  * Anti-Inflammatory drugs
  * Lipid lowering drugs including statins
  * Anti-hypertensive drugs
  * Anti-coagulant drugs
* Body Mass Index (BMI) greater than or equal to 40.
* Pregnant or Lactating
* Inability to communicate effectively with study personnel

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2007-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in inflammatory markers (MCP-1, IL-6, and sICAM-1) at 8 weeks. | Baseline and 8 weeks
  Change was calculated as the value at 8 weeks minus the value at baseline

SECONDARY OUTCOMES:
Change from baseline in red blood cells (RBC) Fatty Acids at 8 weeks. | Baseline and 8 weeks
  Change was calculated as the value at 8 weeks minus the value at baseline
Change from baseline in low-density lipoprotein (LDL) cholesterol at 8 weeks. | Baseline and 8 weeks
  Change was calculated as the value at 8 weeks minus the value at baseline
Change from baseline in high-density lipoprotein (HDL) cholesterol at 8 weeks. | Baseline and 8 weeks
  Change was calculated as the value at 8 weeks minus the value at baseline
Change from baseline in triglycerides at 8 weeks. | Baseline and 8 weeks
  Change was calculated as the value at 8 weeks minus the value at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Gardner, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dewell A, Marvasti FF, Harris WS, Tsao P, Gardner CD. Low- and high-dose plant and marine (n-3) fatty acids do not affect plasma inflammatory markers in adults with metabolic syndrome. J Nutr. 2011 Dec;141(12):2166-71. doi: 10.3945/jn.111.142240. Epub 2011 Oct 26. PMID 22031659
- See also: Study description and summary of results — https://med.stanford.edu/nutrition/research/completed-studies/plant-vs-marine-omega-3s.html